CLINICAL TRIAL: NCT05275673
Title: A Randomized, Open-Label Phase 2 Study of the TORC 1/2 Inhibitor Sapanisertib in Relapsed/Refractory NFE2L2 (NRF2)-Mutated and Wild-Type (WT) Squamous Non-Small Cell Lung Cancer (sqNSCLC)
Brief Title: A Study of Sapanisertib in Relapsed/Refractory NFE2L2-Mutated and Wild-Type Squamous Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision - funding issues
Sponsor: Faeth Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX-228-301
Record Dates: First submitted 2022-02-07; First posted 2022-03-11 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer; Squamous Non-small-cell Lung Cancer; Squamous Non-Small Cell Neoplasm of Lung; NFE2L2 Gene Mutation
Keywords: NSCLC; sqNSCLC; NFE2L2; Next Generation Sequencing; NGS; Mutation; Relapsed; Refractory; Squamous; NRF2; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence; Lung Neoplasms | interventions — sapanisertib

STUDY DESIGN:
Intervention Model Description: 2 dosing schedules: 3 mg once per day (3 mg total) OR 2 mg twice per day (4 mg total)
  Group A: 30 participants randomized 1:1 to one of two dosing schedules
  Group B: approximately 20 participants randomized 1:1 to one of two dosing schedules
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A - NFE2L2 Mutation, Dosing Cohort 1 (Experimental): sapanisertib 3 mg once daily (QD)
  Interventions: Drug: sapanisertib
- Group A - NFE2L2 Mutation, Dosing Cohort 2 (Experimental): sapanisertib 2 mg twice daily (BID)
  Interventions: Drug: sapanisertib
- Group B - NFE2L2 Wild-Type, Dosing Cohort 1 (Experimental): sapanisertib 3 mg QD
  Interventions: Drug: sapanisertib
- Group B - NFE2L2 Wild-Type, Dosing Cohort 2 (Experimental): sapanisertib 2 mg BID
  Interventions: Drug: sapanisertib

INTERVENTIONS:
Drug: sapanisertib — capsules for oral administration
  Other Names: CB-228

SUMMARY:
This is a multicenter, randomized, open-label Phase 2 study of sapanisertib in biomarker-defined populations of sqNSCLC. Patients with NFE2L2 (the name for gene encoding the protein called NRF2)-mutated or wild-type sqNSCLC should have disease that has progressed on or after at least two prior systemic therapies for metastatic disease including platinum-doublet chemotherapy and a programmed cell death 1 ligand 1 (PD-L1) inhibitor. The study will evaluate sapanisertib monotherapy in patients with relapsed/refractory sqNSCLC as two separate groups: Group A: NFE2L2-mutated sqNSCLC and Group B: NFE2L2-WT sqNSCLC.

DETAILED DESCRIPTION:
NFE2L2 mutation status for all patients will be identified using local or central next generation sequencing (NGS) testing on archival or fresh tissue or circulating tumor deoxyribonucleic acid (ctDNA), the results of which must be reviewed and approved by the Sponsor prior to enrollment. Each group will be randomized 1:1 to one of two doses/schedules of sapanisertib. Approximately 30 NFE2L2-mutant and 20 NFE2L2-wild type patients will be enrolled. Patients will be treated with sapanisertib until disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), unacceptable toxicity, withdrawal of consent, or death.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV squamous NSCLC.
* Disease progression during or after prior systemic therapy for metastatic disease, which must include platinum-doublet chemotherapy and immune checkpoint inhibitor therapy (anti-PD-(L)1 +/-anti-CTLA-4), if approved and available, administered as separate lines of therapy or in combination.
* Has study-eligible mutation in NFE2L2 or wild-type NFE2L2 using NGS from a College of American Pathologists- (CAP)-accredited and/or a Clinical Laboratory Improvement Amendments- (CLIA)-certified laboratory
* Must have at least one radiographically measurable lesion per RECIST v1.1 defined as a lesion that is ≥ 10 mm in longest diameter or lymph node that is ≥ 15 mm in short axis imaged by computerized tomography (CT) scan or Magnetic Resonance Imaging (MRI).
* Target lesions situated in a previously irradiated area may be considered measurable if progression has been demonstrated subsequent to radiation therapy.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Adequate Organ Function Laboratory Findings: Absolute neutrophil count (ANC): ≥1,500/mm3, Hemoglobin: ≥9.0 g/dL * Transfusions and growth factors must not be used within 2 weeks prior to randomization to meet these requirements, Platelets: ≥ 100,000/mm3, Calculated creatinine clearance (CrCl): ≥ 40mL/min, Serum total bilirubin: ≤ 1.5× upper limit of normal (ULN) OR ≤ 3 mg/dL for patients with Gilbert's disease, AST (SGOT) and ALT (SGPT): ≤ 2.5× ULN OR ≤ 5× ULN for patients with liver metastases, Fasting triglycerides: < 300 mg/dL, Fasting serum glucose: <160 mg/dL
* A female patient of childbearing potential must:

  1. Have a negative serum or urine pregnancy test within 7 days prior to the first dose of study treatment
  2. Agree to use acceptable methods of contraception(See Section 8.1.2) during the study and for a minimum of 14 days following the last dose of sapanisertib
  3. Post-menopausal females (no menses for >1 year without an alternative medical cause) and surgically sterilized females are exempt from these requirements.
* Male patients must use an effective barrier method of contraception if sexually active with a female of childbearing potential and refrain from donating sperm during the study and for a minimum of 14 days following the last dose of sapanisertib.

Exclusion Criteria:

* Non-squamous cell histology and mixed histology tumors with any small-cell/neuroendocrine component.
* Prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment per investigator's discretion.
* Receipt before the first dose of study drug of any of the following:

  i. Any investigational agent within 4 weeks. ii. Chemotherapy with 3 weeks (6 weeks for nitrosoureas or mitomycin C) iii. Any radiotherapy within 2 weeks prior to randomization with the exception of palliative radiotherapy for isolated tumor lesions
* Major surgery or other anticancer therapy not previously specified within 4 weeks.
* Unable or unwilling to discontinue proton pump inhibitor (PPI) use ≥ 5 days prior to randomization.
* Interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoid treatment.
* Any condition including social, psychiatric or medical (including uncontrolled significant concurrent illness) that in the opinion of the Investigator could interfere with treatment or protocol-related procedures.
* Patients who are pregnant or lactating.
* Symptomatic ascites or pleural effusion. Exception: Patients who are clinically stable following treatment for these conditions (including therapeutic thoraco-or paracentesis) are eligible.
* Refractory nausea and vomiting, uncontrolled diarrhea, malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes or other situation that may preclude adequate absorption of oral study medication.
* Infection requiring more than 5 days of parenteral antibiotics, antivirals, or antifungals within two weeks prior to randomization.
* Patients receiving systemic corticosteroids greater than prednisone 10 mg or equivalent (excluding inhalers or low-dose hormone replacement therapy) within the 7 days before treatment initiation.
* Previous intolerance to mammalian target of rapamycin (mTOR), AKT, or dual PI3K/mTOR inhibitors.
* Patients with symptomatic, active/untreated central nervous system metastasis and/or leptomeningeal disease are not eligible.
* Significant active cardiovascular disease
* Participants who are known to be HIV-positive, unless assessed to be healthy with a low risk of AIDS-related outcomes.
* Known active Hepatitis B or C infection.
* Manifestations of malabsorption due to prior gastrointestinal (GI) surgery, GI disease, or for an unknown reason that may alter the absorption of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Paik, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (14):
- United States (14):
  - UC Davis Comprehensive Cancer Center, Davis, California
  - Providence Medical Group Santa Rosa - Cancer Center, Santa Rosa, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Norton Cancer Institute, Downtown, Louisville, Kentucky
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University - Patient Care Coordinator Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - Thoracic, New York, New York
  - Zangmeister Cancer Center, Columbus, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialist, PC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the individual participant data with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was discontinued on 24 Jan 2023 due to limitations in resources. Of approximately 64 participants planned for the study, 7 participants (11%) were enrolled.
Groups:
- Sapanisertib 3 mg QD: Sapanisertib 3 mg once daily (QD)
- Sapanisertib 2 mg BID: Sapanisertib 2 mg twice daily (BID)
Period: Overall Study
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Study Termination by Sponsor | 2 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Sapanisertib 3 mg QD: Sapanisertib 3 mg orally daily
- Sapanisertib 2 mg BID: Sapanisertib 2 mg orally twice daily
- Total: Total of all reporting groups
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 6
  Black | 1 | 0 | 1
  Unknown | 0 | 0 | 0
NFE2L2 Status [Count of Participants; unit: Participants] — NFE2L2 is the name for a gene encoding the protein called NRF2 in squamous non-small cell lung cancer (sqNSCLC). Participants were enrolled with either NFE2L2-mutated of NFE2L2 wild-type (WT) sqNSCLC.
  Participants
    Participants with NFE2L2-mutated sqNSCLC | 2 | 1 | 3
    Participants with NFE2L2-wild type (WT) sqNSCLC | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Investigator-Assessed Overall Response Rate (ORR) Per RECIST v1.1.
Description: ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) according to the RECIST v1.1 criteria as assessed by the investigator.
Time Frame: 36 months
Population: No data were collected. No evaluation of efficacy endpoints was performed for this early terminated study, as no participant was enrolled for the planned 36 months.
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs, and Deaths
Description: An adverse event (AE) is defined as any untoward, undesired, or unplanned medical occurrence in a patient administered a medicinal product whether or not considered drug related. A serious adverse event (SAE) is defined as an AE that occurs after receiving study treatment (or after signing informed consent and before receiving study treatment if due to a protocol-mandated procedure) that either results in death, is life-threatening, requires inpatient hospitalization, results in persistent or significant disability, results in congenital anomaly or birth defect, or otherwise meets criteria as an important medical event. Events were categorized as related or not related to study drug, and event severity was graded as mild (1), moderate (2), severe (3), life-threatening (4), or fatal (5).
Time Frame: From the first dose through 28 days after the last dose of sapanisertib (up to a maximum of 124 days).
Measure: Count of Participants; unit: Participants
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
Number analyzed (Participants) | 4 | 3
Participants
  AE | 3 | 2
  AE >= Grade 3 | 1 | 1
  Serious AE | 1 | 1
  AE Related to Study Drug | 3 | 1
  Death | 1 | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR is the time between the first documentation of partial response (PR) or a complete response (CR) to the first documentation of progressive disease or death, whichever occurs first.
Time Frame: 36 months
Population: No data were collected. There was no evaluation of efficacy endpoints performed for this early terminated study, as no participant was enrolled for the planned 36 months.
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression as determined by the investigator using RECIST v1.1 or death from any cause, whichever occurs first.
Time Frame: 36 months
Population: as for outcome 3
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS) at 6 and 12 Months
Description: OS is defined as the time from randomization to death due to any cause.
Time Frame: Months 6 and 12
Population: No data were collected. There was no evaluation of efficacy endpoints performed for this early terminated study, as no participant was enrolled for >/= 6 months.
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From enrollment (all-cause mortality) or from the first dose of study drug (adverse events) through the last day on study (up to a maximum of 124 days).
Arm/Group | Sapanisertib 3 mg QD | Sapanisertib 2 mg BID
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/3
Other Adverse Events (participants affected / at risk) | 3/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapanisertib 3 mg QD (N=4) | Sapanisertib 2 mg BID (N=3)
Sepsis (Infections and infestations) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapanisertib 3 mg QD (N=4) | Sapanisertib 2 mg BID (N=3)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by the PI before either a multi-site publication or 18 months after final multi-site study report. PI can only publish their own results and provide 45 days in advance notice. PI must delete any Calithera confidential information from the publication other than study results and give good faith consideration to other comments made by Calithera. The PI must delay the publication for up to 45 days if requested by Calithera and publicly acknowledge Calithera and Pfizer support.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT05275673/Prot_SAP_002.pdf